CLINICAL TRIAL: NCT02066428
Title: A Phase I Randomized Placebo-Controlled, Double-Blind Study to Evaluate Safety and Immunogenicity of AERAS-404 Administered as Different Amounts of Antigen and Adjuvant Combinations in HIV-Negative BCG-Vaccinated Adults Without Evidence of Tuberculosis Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aeras (Other)
Collaborators: Statens Serum Institut (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C-005-404
Record Dates: First submitted 2014-02-17; First posted 2014-02-19 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Tuberculosis
Keywords: BCG Vaccinated; HIV Negative
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- AERAS-404(50mcg H4/0nmol IC31) or Placebo (Experimental): 1 dose
  Interventions: Biological: AERAS-404; Biological: Placebo
- AERAS404 (50mcgH4/100nmol IC31) or Placebo (Experimental): 1 dose
  Interventions: Biological: AERAS-404; Biological: Placebo
- AERAS404 (50mcgH4/0nmol IC31) or Placebo (Experimental): 2 dose
  Interventions: Biological: AERAS-404; Biological: Placebo
- AERAS404 (150mcgH4/0nmol IC31) or Placebo (Experimental): 1 dose
  Interventions: Biological: AERAS-404; Biological: Placebo
- AERAS404 (50mcgH4/5000nmol IC31) or Placebo (Experimental): 1 dose
  Interventions: Biological: AERAS-404; Biological: Placebo
- AERAS404 (50mcgH4/500nmol IC31) or Placebo (Experimental): 2 dose
  Interventions: Biological: AERAS-404; Biological: Placebo
- AERAS404 (Experimental): 2 dose placebo
  Interventions: Biological: Placebo
- AERAS404 (50mcg H4/100nmol IC31) or Placebo (Experimental): 2 dose
  Interventions: Biological: AERAS-404; Biological: Placebo

INTERVENTIONS:
Biological: AERAS-404 — AERAS 404 (H4:IC31) contains a fusion protein of 2 mycobacterial antigens (Ag85B and TB 10.4) formulated in IC31 adjuvant.
  Other Names: H4
  Arms: AERAS-404(50mcg H4/0nmol IC31) or Placebo; AERAS404 (150mcgH4/0nmol IC31) or Placebo; AERAS404 (50mcg H4/100nmol IC31) or Placebo; AERAS404 (50mcgH4/0nmol IC31) or Placebo; AERAS404 (50mcgH4/100nmol IC31) or Placebo; AERAS404 (50mcgH4/5000nmol IC31) or Placebo; AERAS404 (50mcgH4/500nmol IC31) or Placebo
Biological: Placebo — Tris buffer saline consisting (10mM Tris and 169mM NaCI at pH7.4)
  Other Names: Tris Buffered saline

SUMMARY:
Phase I, randomized, double blinded, Placebo-controlled, immunogenicity and dose-range finding study of AERAS-404 in Bacille Calmette-Guerin (BCG) healthy adult male and sterile females.

DETAILED DESCRIPTION:
This ia a Phase I, randomized, placebo-controlled, double-blind study in three groups of healthy adult males or sterile females who are BCG-vaccinated, HIV-negative, and have no evidence of tuberculosis infection.

Sixty-four subjects assigned to one of eight treatment groups to receive one of four different antigen/adjuvant combinations of study vaccine, or placebo control. Within each study group, subjects will be randomized to receive either a single-dose antigen/adjuvant regimen of study vaccine (vaccination with study vaccine on Study Day 0 followed by vaccination with placebo control on Study Day 56) or a two-dose antigen/adjuvant regimen of study vaccine (vaccination with study vaccine on Study Days 0 and 56).

All subjects will be followed for safety and immunogenicity evaluations for 182 days.

The sample sizes specified for each study group were selected because they are judged to be adequate for preliminary safety and immunogenicity evaluations for a Phase I study rather than for statistical reasons. If no SAE are observed among 56 subjects receiving active study vaccine, an approximation to the upper 95% confidence bound on the rate of SAE occurrence would be 5.4%.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Age 18 through 50 years on Study Day 0
3. Completed wriiten Informed Consent
4. BCG vaccination at least 5 years ago,
5. General good health, confirmed by medical history
6. (BMI) between 19 and 33 (kg/m2)
7. Has ability to complete follow-up period of 182 days as required
8. Females must be physically incapable of conception
9. Avoiding elective surgery for the duration of the study
10. Stay in contact with the investigative site for the duration of the study
11. Complete simultaneous enrollment in Aeras Vaccine Development Registry protocol

Exclusion Criteria:

1. Acute illness on the day of randomization
2. Oral temperature >=37.5 degree Celcius on the day of randomization
3. Evidence of significant active infection
4. Used immunosuppressive medication within 42 days before entry into the study
5. Received immunoglobulin or blood products within 42 days before entry into the study
6. Received any investigational drug therapy or investigational vaccine within 182 days
7. Received inactivated influenza vaccine or inactivated tick-borne encephalitis vaccine within 14 days before entry into the study.
8. Current chronic drug therapy including hormone replacement such as thyroxin, insulin, etc.
9. History or laboratory evidence of any past, present or future possible immunodeficiency state which will include any laboratory indication of virus type 1 (HIV-1) infection
10. History of allergic disease or reactions, including eczema.
11. Previous medical history that may compromise safety of subject
12. Evidence of new acute illness that may compromise safety of subject
13. Evidence of chronic hepatitis
14. Inability to discontinue daily medication except contraception
15. History of alcohol or drug abuse within 2yrs
16. Tobacco or cannabis smoking three
17. Positive urine test for illicit drugs
18. History or evidence of any systemic disease on physical examination
19. History of active TB
20. Shared residence within 1 year with an individual on anti-TB treatment
21. All females: nursing
22. Abnormal hemoglobin,hematocrit etc drawn within 36 hours prior to randomization
23. Laboratory test evidence of Mtb infection
24. History of positive tuberculin skin test within past 10 years
25. Received a tuberculin skin test within 3 years
26. History of autoimmune disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2007-11; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of one or two injections of two AERAS 404 antigen amounts administered with three different amounts of adjuvant | All subjects will be followed for safety and immunogenicity evaluations for 182 days. A total of eleven clinic visits are planned (excluding screening) for all subjects
  Serious adverse events (SAE) will be collected on subjects throughout their participation in the study. Solicited and unsolicited AEs will be collected through 28 days after each vaccination.The safety profile of the different antigen/adjuvant treatment regimens will be described. Listings will be provided for all subjects with serious adverse events (SAE). All adverse events and clinically relevant laboratory results will be summarized across time points to examine the relationship between treatment regimens (i.e., number of doses and level of antigen/adjuvant) and key safety endpoints including number (percentage) of solicited and spontaneous adverse events and number (percentage) of subjects with newly abnormal post-vaccination laboratory values based on predefined toxicity criteria. Adverse events will also be summarized by severity and relationship to study vaccine by treatment regimen.

SECONDARY OUTCOMES:
Evaluate the immunogenicity of one or two injections of two AERAS 404 antigen amounts administered with three different amounts of adjuvant. | all subjects will have immunology samples taken at 9 time points over 182 days
  Assessment of immune response will be based on the percentage of CD4 and CD8 T cells producing any of three cytokines (interferon gamma, IFN-γ; tumor necrosis factor alpha, TNF-α; and/or interleukin-2, IL-2) or any combination of these three cytokines simultaneously in response to stimulation with two the antigenic peptide pools contains 85B and TB10.4 representing the entire amino acid sequences of mycobacterial antigens Ag85B and TB10.4, respectively. Responses will be measured by flow cytometry using a qualified intracellular cytokine staining (ICS) assay

CONTACTS AND LOCATIONS:
Overall Officials: Zhongkai SHI, MD, Study Director — Aeras; Jan Andersson, MD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Karolinska University Hospital, Huddinge, Stockholm County, Sweden

REFERENCES:
- [Derived] Norrby M, Vesikari T, Lindqvist L, Maeurer M, Ahmed R, Mahdavifar S, Bennett S, McClain JB, Shepherd BM, Li D, Hokey DA, Kromann I, Hoff ST, Andersen P, de Visser AW, Joosten SA, Ottenhoff THM, Andersson J, Brighenti S. Safety and immunogenicity of the novel H4:IC31 tuberculosis vaccine candidate in BCG-vaccinated adults: Two phase I dose escalation trials. Vaccine. 2017 Mar 14;35(12):1652-1661. doi: 10.1016/j.vaccine.2017.01.055. Epub 2017 Feb 17. PMID 28216183